CLINICAL TRIAL: NCT03943784
Title: Endoscopic Variceal Ligation as Primary Prophylaxis for Upper Gastrointestinal Bleeding in Children
Brief Title: Endoscopic Variceal Ligation in Children
Status: Completed | Type: Observational
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Jesús Quintero, Responsible of Pediatric Hepatology and Liver Transplant Department, Hospital Vall d'Hebron
Other Study IDs: 31/2019
Record Dates: First submitted 2019-05-03; First posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Esophageal Varices in Cirrhosis of the Liver; Upper Gastrointestinal Bleeding; Endoscopy; Child
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Propranolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic Variceal Ligation: From January 2014 to April 2017, all paediatric patients with a known chronic liver disease with suspicion of portal hypertension who presented grade 2 or 3 esophageal varices or red spots in the upper endoscopy received primary prophylaxis with endoscopic variceal ligation.
  Interventions: Procedure: Endoscopic Variceal Ligation
- Propranolol Group: Patients in the Endoscopic Variceal Ligation group were compared with an historical cohort of 30 consecutive patients with portal hypertension and grade 2 or 3 esophageal varices or red spots who received propranolol as primary prophylaxis from January 2009 to December 2013. All patients were treatment-naïve in regards of their upper gastrointestinal bleeding prophylaxis at the time of the first upper endoscopy.
  Interventions: Drug: Non-Selective Beta-Blocking Agent

INTERVENTIONS:
Procedure: Endoscopic Variceal Ligation — Endoscopic varices ligation was performed with a six-shooter multiband ligator (Cook Medical, Limerick, Ireland) if medium to large varices or reddish spots, regardless of the grade of the varix, were observed. Each varix was ligated 1-2 cm above the gastro-esophageal junction, with 1 or 2 rubber bands and using no more than 5 rubber bands per session.
  Groups: Endoscopic Variceal Ligation
Drug: Non-Selective Beta-Blocking Agent — Patients of the Propranolol group that presented medium to large esophageal varices without contraindication to Non-Selective Beta-Blockers, received propranolol, 1 mg/Kg/day every 8 hours, titrated to reduce the basal heart rate in 25% and not exceeding 5 mg/Kg/day. Patients were evaluated monthly until this reduction in heart rate was achieved, and every three to six months thereafter.
  Other Names: Propranolol
  Groups: Propranolol Group

SUMMARY:
This is an ambispective single-center cohort study of pediatric patients with portal hypertension and esophageal varices. The study was designed to evaluate the efficacy and safety of primary prophylaxis with endoscopic variceal ligation to prevent upper gastrointestinal bleeding compared to non-selected beta-blockers prophylaxis.

DETAILED DESCRIPTION:
Endoscopic Variceal Ligation group; Inclusion criteria From January 2014 to April 2017, a study group was created, including all paediatric patients with a known chronic liver disease with suspicion of portal hypertension and grade 2 or 3 OV or red spots, regardless of the grade of the OV diagnosed by endoscopy.

Propanolol group Patients in the Endoscopic Variceal Ligation study group were compared with an historical cohort of 30 consecutive patients with portal hypertension and grade 2 or 3 esophageal varices or red spots, regardless of the grade of the esophageal varices in the upper endoscopy, who received propranolol as primary prophylaxis from January 2009 to December 2013.

Ligation sessions were performed every 6 weeks until varices eradication. When eradication was achieved, upper endoscopy was performed at 2 and 6 months to assess the efficacy of the treatment. If no varices were observed, upper endoscopies were performed once a year thereafter.

Eradication was defined as disappearance of all varices or reduction to grade 1 small varices without reddish spots and no gastric varices.

ELIGIBILITY:
Inclusion Criteria for endoscopic variceal ligation cohort

* All paediatric patients (< 18 years)
* Known chronic liver disease
* Suspicion of portal hypertension based on splenomegaly in the ultrasound, presence of collaterals in the abdominal wall or low platelet count (<150.000 platelets/L),
* Grade 2 or 3 esophageal varices or red spots, regardless of the grade of the esophageal varices diagnosed by endoscopy
* From January 2014 to April 2017

Exclusion Criteria for endoscopic variceal ligation cohort:

* Patients initially treated with Non-selective beta blockers and subsequently treated with endoscopic variceal ligation as primary prophylaxis were excluded of the study.
* Patients for whom endoscopic variceal ligation was not feasible because of patients' weight/seize were also excluded of the study.

Inclusion Criteria for propranolol cohort

* All paediatric patients (< 18 years)
* Known chronic liver disease
* Suspicion of portal hypertension based on splenomegaly in the ultrasound, presence of collaterals in the abdominal wall or low platelet count (<150.000 platelets/L),
* Grade 2 or 3 esophageal varices or red spots, regardless of the grade of the esophageal varices diagnosed by endoscopy
* That received propranolol as primary prophylaxis
* From January 2009 to December 2013.

Exclusion Criteria propranolol cohort:

* Patients initially treated with non-selective beta blockers and subsequently treated with endoscopic variceal ligation as primary prophylaxis were excluded of the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All pediatric patients with a known chronic liver disease with suspicion of portal hypertension who presented grade 2 or 3 esophageal varices or red spots, regardless of the grade of the esophageal varices diagnosed by endoscopy from January 2009 to April 2017 that received propranolol or endoscopic variceal ligation as a primary prophylaxis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Number of patients that present the first episode of Upper Gastrointestinal Bleeding after the use of endoscopic variceal ligation as a prophylactic treatment (Efficacy) | From the moment the patients received the endoscpoic variceal ligation to the end of the follow-up (April 2019)
  From the moment that the endoscopic variceal ligation was performed, the number of patients that present the first episode of upper gastrointestinal bleeding due to esophageal varices will be recorded
Number of patients that present adverse events related to the use of endoscopic variceal ligation as a prophylactic treatment (Safety) | From the moment the patients received the endoscpoic variceal ligation to the end of the follow-up (April 2019)
  Hematology and biochemistry parameters and adverse events notified during the study will be recorded in order to evaluate the safety and tolerability of endoscopic variceal ligation as prophylactic treatment of upper gastrointestinal bleeding in pediatric patients

SECONDARY OUTCOMES:
Survival at 1 year after prophylactic treatment (endoscopic or propranolol) | Survival will be reported at 1 year after the start of the prophylactic treatment
  Survival was defined as the time from endoscopic variceal ligation/propranolol start to death due to upper gastrointestinbal bleeding or date of last follow-up, measured in months
Survival at 3 year after prophylactic treatment (endoscopic or propranolol) | Survival will be reported at 3 years after the start of the prophylactic treatment
  Survival was defined as the time from endoscopic variceal ligation/propranolol start to death due to upper gastrointestinbal bleeding or date of last follow-up, measured in months
Transplant-free survival at 1 year | Transplant-free survival wil be reported at 1 year after the start of the prophylactic treatment
  Transplant-free survival was defined as the time from endoscopic variceal ligation or propranolol start to the date of transplantation, measured in months
Transplant-free survival at 3 years | Transplant-free survival wil be reported at years after the endoscopic prophylaxis
  Transplant-free survival was defined as the time from endoscopic variceal ligation or propranolol star to the date of transplantation, measured in months
Esophageal varices eradication with endoscopic treatment | From the first episode of variceal ligation to eradication
  The number of patients that present esophageal varices eradication using endoscopic variceal ligation. Eradication was defined as disappearance of all varices or reduction to grade 1 small varices without reddish spots and no gastric varices.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quintero J, Juamperez J, Mercadal-Hally M, King ML, Ortega J, Molino JA, Abu-Suboh M, Dot J, Nuno R, Montferrer N, Armengol JR, Charco R. Endoscopic variceal ligation as primary prophylaxis for upper GI bleeding in children. Gastrointest Endosc. 2020 Aug;92(2):269-275. doi: 10.1016/j.gie.2020.02.035. Epub 2020 Feb 29. PMID 32119939